CLINICAL TRIAL: NCT04751929
Title: A Phase II Multi-Center Trial of Abemaciclib With or Without Atezolizumab in Metastatic Castration Resistant Prostate Cancer
Brief Title: Abemaciclib With or Without Atezolizumab for mCRPC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Atish Choudhury, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-701
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Abemaciclib; Atezolizumab; CDK4/6; Immunotherapy; PD-L1
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abemaciclib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Biomarker-Unselected Abemaciclib Monotherapy (Randomized) (Experimental): Participants in the Biomarker-Unselected Cohort, defined as those whose tumors are not known to have mutations in the CDK12 gene will be randomized to either receive Abemaciclib as monotherapy or in combination with Atezolizumab
  * Monotherapy : Participants will receive Abemaciclib orally 2x daily
  Interventions: Drug: Abemaciclib
- Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) (Experimental): Participants in the Biomarker-Unselected Cohort, defined as those whose tumors are not known to have mutations in the CDK12 gene will be randomized to either receive Abemaciclib as monotherapy or in combination with Atezolizumab
  * Combination Therapy: Participants will receive Abemaciclib orally 2x daily and Atezolizumab intravenously Day 1 of each 21-Day cycle
  Interventions: Drug: Abemaciclib; Drug: Atezolizumab
- CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) (Experimental): Participants in the CDK12 Mutation Cohort defined as those whose tumors are known to have mutations in the CDK12 gene are not randomized but are assigned to receive either Atezolizumab monotherapy or in combination with Abemaciclib based on how many participants in this cohort previously received study treatment.
  Atezolizumab monotherapy will be given to participants 1-5, these participants will receive Atezolizumab intravenously Day 1 of each 21-Day cycle
  Interventions: Drug: Atezolizumab
- CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) (Experimental): Participants in the CDK12 Mutation Cohort defined as those whose tumors are known to have mutations in the CDK12 gene are not randomized but are assigned to receive either Atezolizumab monotherapy or in combination with Abemaciclib based on how many participants in this cohort previously received study treatment.
  Combination Therapy will be given to participants 6-21, these participants will receive Abemaciclib orally 2x daily and Atezolizumab intravenously Day 1 of each 21-Day cycle
  Interventions: Drug: Abemaciclib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Abemaciclib — Taken orally 2x daily
  Other Names: Verzenio
  Arms: Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized); Biomarker-Unselected Abemaciclib Monotherapy (Randomized); CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
Drug: Atezolizumab — Intravenously Day 1 of 21 day cycle
  Other Names: Tecentriq
  Arms: Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized); CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized); CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized)

SUMMARY:
This trial is testing whether a molecularly targeted chemotherapy drug called abemaciclib and an immunotherapy drug called atezolizumab, alone or in combination, are effective in shrinking or preventing the growth of metastatic prostate cancer. The trial is also testing the safety of the combination of abemaciclib with atezolizumab.

DETAILED DESCRIPTION:
This is a multi-center, open label Phase II study of patients with metastatic castration resistant prostate cancer (mCRPC) who will be treated with abemaciclib and atezolizumab alone or in combination.

The U.S. Food and Drug Administration (FDA) has not approved abemaciclib or atezolizumab alone or in combination for use in prostate cancer. Abemaciclib is an orally administered molecularly targeted chemotherapy drug called a cyclin-dependent kinase inhibitor, which acts to block the ability of cancer cells to divide and thus prevents tumors from growing. In the laboratory setting, this drug is effective in prostate cancer models that have become resistant to standard hormonal treatments, and this drug is currently being studied for its effectiveness in prostate cancer in other clinical trials. Atezolizumab is an intravenously administered drug called an immune checkpoint inhibitor, which acts to activate the immune system to kill cancer cells. Atezolizumab is ineffective on its own in most patients with prostate cancer, but is being tested in combination with other drugs for prostate cancer in other clinical trials. Multiple research groups have demonstrated in laboratory model systems that abemaciclib can may make immune checkpoint inhibitors more effective.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

The study design divides study participants into two separate cohorts. The first cohort is a set of subjects whose tumors are not known to have mutations in the CDK12 gene (the "biomarker unselected cohort") - either because tumor tissue never underwent genetic profiling, or because genetic profiling was performed but did not demonstrate a mutation in the CDK12 gene. In this "biomarker unselected cohort," this study will be testing whether abemaciclib alone or in combination with atezolizumab is an effective treatment strategy.

The second cohort of participants is a set of subjects whose tumors are known to have mutations in the CDK12 gene based on genetic profiling of the tumor that occurred prior to enrollment on this study. Prior studies suggest that cancers with mutations in the CDK12 gene can shrink in response to immune checkpoint inhibitors. This study will be testing in study participants whose tumors are known to have mutations in CDK12 whether atezolizumab alone or in combination with abemaciclib is an effective treatment strategy.

In addition, the trial is testing the safety of the combination of the two drugs in both cohorts.

Participants will receive study treatment for as long as they do not have serious side effects and their disease does not get worse. Participants will be followed after completion of study treatment for up to 24 months

It is expected that about 75 people will take part in this research study.

Eli Lilly and Company is supporting this research study by providing funding for research and the study drug abemaciclib. Genentech, Inc. is supporting the study by providing the study drug atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic castration resistant prostate cancer (mCRPC), with histologic confirmation of adenocarcinoma of the prostate (without evidence of small cell carcinoma), with progressive disease at the time of study entry by either

  * Sequence of at least 2 rising PSA values at a minimum of 1-week intervals
  * Radiographic progression per RECIST1.1 for soft tissue and/or per PCWG3 for bone, with or without PSA progression
* Adult males 18 years of age or older.
* ECOG performance status of 0 or 1
* Patients must have metastatic disease by bone scintigraphy or other nodal or visceral lesions on CT or MRI with a bone or soft tissue lesion amenable to image-guided percutaneous biopsy, and the patient must be evaluable for disease response by either

  * Baseline PSA ≥ 2.0 ng/mL OR
  * Measurable disease per RECIST 1.1
* Past progression or intolerance to at least one novel antiandrogen therapy (abiraterone, enzalutamide, galeterone, apalutamide, darolutamide, orteronel, seviteronel or equivalent) in either the hormone-sensitive or castration-resistant disease setting.
* Not a candidate for docetaxel or cabazitaxel chemotherapy due to:

  * progression within 12 months of completion or intolerance to prior taxane OR
  * refusal of taxane OR
  * contraindication to, or lack of fitness for taxane OR
  * Investigator assessment that taxane is not clinically indicated or preferred.
* Maintenance of castration status, defined as serum testosterone level of less than 50 ng/dL. Patients must be surgically castrate or maintained on LHRH agonist or antagonist therapy for the duration of the study period.
* Must have recovered from any treatment-related toxicities to ≤ CTCAE grade 1.

  * Patients with ≤ CTCAE grade 2 anorexia, alopecia, neuropathy, and/or fatigue however, are also permitted to enroll.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * hemoglobin ≥9 g/dL (without transfusion or growth factor in prior 28 days)
  * platelets ≥100,000/mcL (without transfusion or growth factor in prior 28 days)
  * total bilirubin ≤1.5 × institutional upper limit of normal, unless the subject has known or suspected Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤1.5 × institutional upper limit of normal
  * creatinine clearance ≥30 mL/min/1.73 m2
* Life expectancy of at least 6 months, as determined by a study Investigator.
* Ability to swallow oral medications.
* Ability to understand and willingness to sign an IRB-approved informed consent.
* Additional Inclusion Criteria (Arm C patients)

  * Must have documentation (via CLIA approved, CAP certified next generation sequencing [NGS] assay report) of genomic aberration resulting in CDK12 loss of function in metastatic tumor tissue.

    * Patients whose tumors have not previously undergone NGS are not eligible for Arm C but are eligible for the randomized unselected cohorts.

Exclusion Criteria:

* Clinical evidence of, or known and untreated metastatic CNS disease.
* Concurrent active malignancy.

  * Patients with non-melanomatous skin cancer, cancer not needing active therapy for at least 2 years, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are also permitted to enroll.
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to planned cycle 1 day 1 of study treatment.
* Patients who have received oral anti-neoplastic intervention such as an oral hormonal agent, PARP inhibitor, AR targeted therapy, or oral experimental agent within 14 days prior to planned cycle 1 day 1 of study treatment.
* Prior treatment with an inhibitor of CDK4 and/or 6.
* Prior treatment with an inhibitor of PD-1, PD-L1, or PD-L2.
* Patients on concurrent therapy with a moderate or strong CYP3A4 inducer or inhibitor which cannot be safely stopped at least five half-lives prior to initiation of therapy with abemaciclib.
* Evidence of an active autoimmune disease that has required systemic treatment within the last 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

  * Patients with conditions requiring replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are permitted to enroll.
* Live vaccine within 30 days of registration.
* Active smoking or a history of smoking greater than 20 pack-years (i.e. # packs of cigarettes smoked per day × # of years patient has smoked > 20).
* Prior history of radiation therapy to thorax (including to lungs/pleura, esophagus, intrathoracic lymph nodes, C7-L2 vertebrae, or ribs) for any reason and any duration/dose.
* Any history of interstitial lung disease, pneumonitis or idiopathic pulmonary fibrosis, regardless of remission or immunosuppression status.
* Any history of lung cancer, regardless of stage or treatment
* Any of the following abnormalities on pre-treatment pulmonary function testing:

  * FEV1/FVC < lower limit of normal (LLN) and FEV1 < 75% predicted OR
  * FVC < 70% of predicted, regardless of FEV1/FVC ratio OR
  * DLCO (corrected for hemoglobin) < 70% of predicted
* Active bacterial or fungal infection, or known detectable viral infection (e.g., Human Immunodeficiency Virus [HIV] or viral hepatitis).
* Arterial or venous thromboembolic event within the last 3 months.
* Significant infection, medical condition, or social situation which, in the opinion of the investigator, would preclude participation or limit the patient's ability to comply with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2025-12-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Atish Choudhury, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Biomarker-Unselected Abemaciclib Monotherapy (Randomized): Participants in the Biomarker-Unselected Cohort, defined as those whose tumors are not known to have mutations in the CDK12 gene will be randomized to either receive Abemaciclib as monotherapy or in combination with Atezolizumab
  * Monotherapy : Participants will receive Abemaciclib orally 2x daily
  Abemaciclib: Taken orally 2x daily
- Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized): Participants in the Biomarker-Unselected Cohort, defined as those whose tumors are not known to have mutations in the CDK12 gene will be randomized to either receive Abemaciclib as monotherapy or in combination with Atezolizumab
  * Combination Therapy: Participants will receive Abemaciclib orally 2x daily and Atezolizumab intravenously Day 1 of each 21-Day cycle
  Abemaciclib: Taken orally 2x daily
  Atezolizumab: Intravenously Day 1 of 21 day cycle
- CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized): Participants in the CDK12 Mutation Cohort defined as those whose tumors are known to have mutations in the CDK12 gene are not randomized but are assigned to receive either Atezolizumab monotherapy or in combination with Abemaciclib based on how many participants in this cohort previously received study treatment.
  Atezolizumab monotherapy will be given to participants 1-5, these participants will receive Atezolizumab intravenously Day 1 of each 21-Day cycle
  Atezolizumab: Intravenously Day 1 of 21 day cycle
- CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized): Participants in the CDK12 Mutation Cohort defined as those whose tumors are known to have mutations in the CDK12 gene are not randomized but are assigned to receive either Atezolizumab monotherapy or in combination with Abemaciclib based on how many participants in this cohort previously received study treatment.
  Combination Therapy will be given to participants 6-21, these participants will receive Abemaciclib orally 2x daily and Atezolizumab intravenously Day 1 of each 21-Day cycle
  Abemaciclib: Taken orally 2x daily
  Atezolizumab: Intravenously Day 1 of 21 day cycle
Period: Overall Study
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
Started | 7 | 8 | 4 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 8 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Rising PSA | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Progressive Disease | 3 | 4 | 4 | 0
Not completed — Death | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the Monotherapy (Non-Randomized) or the CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) arms. One patient in each of the following arms, Biomarker-Unselected Abemaciclib Monotherapy (Randomized) and CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized), did not initiate study treatment and was therefore excluded from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) | Total
Number analyzed (Participants) | 7 | 8 | 4 | 0 | 19
Age, Continuous [Median (Full Range); unit: years] | 71 [60 to 77] | 70 [64 to 79] | 69 [62 to 75] |  | 70 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 |  | 0
  Male | 7 | 8 | 4 |  | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 1 | 1 | 0 |  | 2
  White | 6 | 7 | 3 |  | 16
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
ECOG performance status [Count of Participants; unit: Participants]
  0; Fully active, able to carry on all pre-disease activities without restriction (best outcome) | 3 | 6 | 3 |  | 12
  1; Restricted in physically strenuous activity but ambulatory and able to carry out light work | 4 | 2 | 1 |  | 7

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression Free Survival (PFS) Rate
Description: The percentage of participants alive and progression-free at 6 months, as assessed by RECIST 1.1 and PCWG3.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
Number analyzed (Participants) | 7 | 8 | 4 | 0
percentage of participants | 100 [100 to 100] | NA [NA to NA] — The median and its 95% CI have not been reached, as the KM curve has not crossed the 50% point. | 50 [10 to 81] |

2. Primary Outcome: Objective Response Rate (ORR)
Description: The percentage of evaluable patients who had radiographic response (complete response or partial response) by RECIST 1.1 criteria OR 50% decline in PSA from pretreatment baseline per PCWG3 criteria.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
Number analyzed (Participants) | 7 | 8 | 4 | 0
percentage of participants | 0 [0 to 0] | 12.5 [0.6 to 47] | 0 [0 to 0] |

3. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicity (DLT) in Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) and CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) Arms
Description: DLT was assessed by Bayesian Continuous Toxicity Monitoring in Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) and CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) arms.
Time Frame: DLTs were collected while participants on treatment. Treatment duration up to 18 months.
Population: Only for Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) and CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) arms
Measure: Count of Participants; unit: Participants
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
Number analyzed (Participants) | 0 | 8 | 0 | 0
Participants | 0 | 4 | 0 | 0

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Proportion of evaluable patients who had complete response (CR), partial response (PR) or stable disease (SD) as their best response to treatment in arms biomarker-unselected abemaciclib monotherapy (randomized), biomarker-unselected abemaciclib + atezolizumab (randomized), and CDK12 mutation abemaciclib + atezolizumab (non-randomized)
Time Frame: From treatment initiation to end of treatment, with follow-up for up to 2 years after treatment discontinuation
Reporting Status: Not Posted

5. Secondary Outcome: Duration of Response (DOR)
Description: The time from the first documented complete response (CR) or partial response (PR) to the earliest date of disease progression or death, whichever occurs first, as determined by PCWG3 criteria.
Time Frame: From the date of first documented CR or PR until disease progression or death, or up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Duration of Therapy (DOT)
Description: The length of time from the first administration of study treatment to the date of treatment discontinuation for any reason
Time Frame: From treatment initiation until treatment discontinuation for any reason
Reporting Status: Not Posted

7. Secondary Outcome: Time to Progression (TTP)
Description: The duration of time from the first administration of study treatment to the date of first documented disease progression, as determined by Prostate Cancer Working Group 3 (PCWG3) criteria. Patients without documented progression are censored at the last tumor assessment date.
Time Frame: From treatment initiation until documented disease progression, or assessed up to 2 years
Reporting Status: Not Posted

8. Secondary Outcome: 12-month Overall Survival (OS)
Description: The percentage of participants who are alive 12 months after the start of treatment
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
Number analyzed (Participants) | 7 | 8 | 4 | 0
percentage of patients | 83 [39 to 97] | 50 [20 to 74] | 75 [22 to 95] |

9. Secondary Outcome: Number of Participants With Maximum Grade Adverse Events by CTCAE v5.0
Description: Number of participants experiencing adverse events, categorized by the maximum grade according to CTCAE v5.0.
Time Frame: From treatment initiation through 100 days after last dose for treatment-emergent adverse events, and up to 2 years after last dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From treatment initiation through 100 days after last dose for treatment-emergent adverse events, and up to 2 years after last dose. Maximum treatment duration was 18 months.
Description: A serious adverse event is classified using physician's discretion. All adverse events resulting in death, life threatening events, significant disability, prolonged hospitalization, congenital abnormality/birth defect, or new cancer will be considered a serious adverse event.
  No patients were accrued in the CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) arm.
Arm/Group | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized)
All-Cause Mortality (participants affected / at risk) | 5/7 | 7/8 | 4/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/7 | 4/8 | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 6/7 | 8/8 | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) (N=7) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) (N=8) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) (N=4) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0/0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0/0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0/0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0/0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0/0 | 0
Joint infection (Infections and infestations) | 1 | 0 | 0/0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0/0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0/0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0/0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0/0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0/0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0/0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0/0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0/0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0/0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biomarker-Unselected Abemaciclib Monotherapy (Randomized) (N=7) | Biomarker-Unselected Abemaciclib + Atezolizumab (Randomized) (N=8) | CDK12 Mutation Atezolizumab Monotherapy (Non-Randomized) (N=4) | CDK12 Mutation Abemaciclib + Atezolizumab (Non-Randomized) (N=0)
Anemia (Blood and lymphatic system disorders) | 5 | 7 | 4 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 5 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Edema limbs (General disorders) | 0 | 1 | 2 | 0
Fatigue (General disorders) | 2 | 5 | 2 | 0
Fever (General disorders) | 0 | 3 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 0
Alkaline phosphatase increased (Investigations) | 2 | 3 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Cardiac troponin T increased (Investigations) | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 4 | 5 | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 4 | 0 | 0
Platelet count decreased (Investigations) | 4 | 3 | 1 | 0
Weight loss (Investigations) | 1 | 2 | 0 | 0
White blood cell decreased (Investigations) | 3 | 3 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04751929/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT04751929/ICF_001.pdf